CLINICAL TRIAL: NCT02430714
Title: Post-marketing Surveillance of Lenvatinib Mesylate (Lenvima Capsule) in Patients With Unresectable Thyroid Cancer (Study LEN01T)
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: LEN01T
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2018-07

CONDITIONS: Thyroid Neoplasms
Keywords: Thyroid Cancer; Lenvima; Post-marketing surveillance; LEN01T; All-Patient Investigation; Lenvatinib Mesylate
MeSH Terms: conditions — Thyroid Neoplasms | interventions — lenvatinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arm 1: A prospective, centrally registered investigation will be conducted. The new administering participants are to be registered at the time of administration.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — 24mg once daily oral dosing to Unresectable thyroid cancer patients
  Other Names: E7080, Lenvima

SUMMARY:
This study is a post-marketing surveillance of lenvatinib in participants with unresectable thyroid cancer. The objectives of this study are to capture unknown adverse reactions, incidences of adverse drug reaction, efficacy, factors considered to have effect to safety and effectiveness, and incidences of hypertension, hemorrhagic events and thromboembolic event, and liver disorder.

ELIGIBILITY:
Inclusion Criteria:

1. All participants with unresectable thyroid cancer and administrated Lenvatinib.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants with unresectable thyroid cancer and administrated Lenvatinib in Japan
Sampling Method: Non-Probability Sample
Enrollment: 629 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2016-11-06 (Actual); Study Completion 2016-11-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs)/adverse drug reactions (ADRs) | up to 1 year

SECONDARY OUTCOMES:
Overall survival (OS) | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yasunori Megumi, Study Director — Drug Fostering and Evolution Coordination Department, Corporate Medical Affairs Headquarters, Eisai Co., Ltd.
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo